CLINICAL TRIAL: NCT04282551
Title: The Effect of Oligosaccharides Versus a Placebo on Bowel Habits in Children With Functional Constipation
Brief Title: The Inside Study: Oligosaccharides Versus Placebo in Functional Constipation
Acronym: Inside
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University and Research (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); FrieslandCampina, Amersfoort, The Netherlands (Unknown); Sensus (Royal Cosun), the Netherlands. (Unknown)
Responsible Party: Principal Investigator, Clara Belzer, Associate Professor, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL70126.081.19
Record Dates: First submitted 2019-12-06; First posted 2020-02-24 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Functional Constipation
Keywords: oligosaccharides
MeSH Terms: interventions — Diet Therapy; Oligosaccharides

STUDY DESIGN:
Intervention Model Description: Parallel study with three arms of 13 weeks in total per participant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oligosaccharide group 1 (Experimental)
  Interventions: Other: dietary intervention with oligosaccharides
- oligosaccharide group 2 (Experimental)
  Interventions: Other: dietary intervention with oligosaccharides
- placebo group (Placebo Comparator)
  Interventions: Other: dietary intervention with oligosaccharides

INTERVENTIONS:
Other: dietary intervention with oligosaccharides — intervention with oligosaccharide 1 or 2, or placebo, given once a day

SUMMARY:
In the present randomised double blind controlled study, the investigators will study the effects of oligosaccharides vs a placebo on the change in stool consistency and stool frequency in children with functional constipation.

DETAILED DESCRIPTION:
Functional constipation (FC) in children is a common gastrointestinal (GI) disorder with a worldwide prevalence ranging from 0.7% to 29.6%. Complaints include infrequent bowel movement, painful defecation due to hard and/or large stools, fecal incontinence, and abdominal pain. Although the condition is rarely life-threatening, it strongly impairs quality of life. Oligosaccharides have been shown to relieve constipation symptoms in young adults and elderly. However, sufficient evidence is lacking linking oligosaccharides intake to improve symptoms in children with FC. The investigators hypothesize that oligosaccharides might be able to relieve symptoms of constipation in young children as well, among which softening stools.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria, as considered by a medical doctor:

* Written informed consent
* Aged 1-3 years
* Children that meet the Rome IV criteria for functional constipation

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Children who suffer from any other GI complaints than functional constipation, known structural GI abnormalities, or previous GI surgery
* Any condition that would make it unsafe for the child to participate.
* Children with clinically significant cardiac, vascular, liver, pulmonary, psychiatric disorders, severe renal insufficiency, human immunodeficiency virus, acquired immunodeficiency syndrome, hepatitis B or C or known abnormalities of haematology, urinalysis, or blood biochemistry
* Children who are allergic to cow's milk or fish
* Use of antibiotics or other medicines or food supplements, and breast milk-feeding, 4 weeks prior to the study, except for the allowed escape medication
* Children that participate in another clinical trial

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Stool consistency | Stool consistency will be measured at different time points during a study period of 13 weeks.
  Change in stool consistency measured by the a stool questionnaire; 5 points stool scale from 1 hard to 5 watery (modified Bristol Stool Form Scale)

SECONDARY OUTCOMES:
Stool frequency in number of cases (%) | These outcome measures will be measured at different time point during a study period of 13 weeks.
  Stool frequency - number of times a child has stools a day as reported in a diary.
Stool consistency in number of cases (%) | These outcome measures will be measured at different time point during a study period of 13 weeks.
  Stool consistency - % of stools in a certain stool scale score as measured via a 5 point stool scale

CONTACTS AND LOCATIONS:
Overall Officials: Clara Belzer, PhD, Principal Investigator — Wageningen University and Research; Marc A Benninga, PhD, Principal Investigator — Emma Children's Hospital, UMC Amsterdam
Locations (1):
- Emma Children's Hospital, UMC Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wegh CAM, Schoterman MHC, Vaughan EE, van der Zalm SCC, Smidt H, Belzer C, A Benninga M. Effect of prebiotic oligosaccharides on bowel habit and the gut microbiota in children with functional constipation (Inside study): study protocol for a randomised, placebo-controlled, multi-centre trial. Trials. 2024 Apr 5;25(1):238. doi: 10.1186/s13063-024-08050-8. PMID 38576033